CLINICAL TRIAL: NCT02880215
Title: Development of Attention Bias Modification for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christopher G. Beevers, Professor and Director of the Institute for Mental Health Research, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201600258; R33MH109600-01A1 (NIH)
Record Dates: First submitted 2016-08-17; First posted 2016-08-26 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Bias Modification (Experimental): Behavioral intervention designed to improved negative attention bias.
  Interventions: Behavioral: Attention Bias Modification
- Cognitive Control Training (Experimental): Behavioral intervention designed to improve sustained attention.
  Interventions: Behavioral: Cognitive Control Training
- Assessment Only (No Intervention): Assessment only with no active intervention.

INTERVENTIONS:
Behavioral: Attention Bias Modification — Behavioral intervention designed to decrease negative attention bias.
  Arms: Attention Bias Modification
Behavioral: Cognitive Control Training — Behavioral intervention designed to improve sustained attention.
  Arms: Cognitive Control Training

SUMMARY:
Although negatively biased attention has a central theoretical and empirical role in the maintenance of depression, there are few behavioral treatments that successfully target and improve this deficit. The current proposal builds upon prior work and aims to further develop an attention bias modification intervention. The investigators propose to develop a highly specific intervention that directly targets negative attention bias and the neurobiology that supports it, using cutting-edge cognitive neuroscience to inform treatment development and improve quality of life of patients whose psychopathology is maintained by negative attention bias.

DETAILED DESCRIPTION:
The overall goal of this project is to continue development of an attention bias modification (ABM) intervention that targets and reduces negative attention bias among adults with elevated symptoms of depression. The investigators' prior work indicates that attention bias for negative information is associated with the maintenance of depression and that neural circuitry within frontal-parietal brain networks supports biased attention for negative information, thus allowing us to develop specific and targeted interventions that directly alter the neurobiology of negative attention bias. The proposed R33 study builds upon the investigators' prior National Institute of Mental Health (NIMH) funded work (R21MH092430), which examined whether ABM reduces negative attention bias and improves symptoms of depression. Findings indicate that compared to placebo ABM, active ABM reduced negative attention bias and increased resting state connectivity within a neural circuit (i.e., middle frontal gyrus and dorsal anterior cingulate cortex) that supports control over emotional information. Further, change in negative attention bias from pre- to post-ABM was significantly correlated with depression symptom change but only in the active training condition. Importantly, a 40% decrease in symptoms was observed in the active training condition; however, similar symptom reduction was also observed in the "placebo ABM" condition. Exploratory analyses indicated that placebo training may have promoted depression improvement by enhancing sustained attention. Although these preliminary findings are encouraging and demonstrate that ABM successfully alters the treatment target (i.e., negative attention bias), the investigators' prior work is among the first to document efficacy of ABM among adults with clinically significant depression. It is now prudent and necessary to obtain additional efficacy evidence for ABM before moving forward with large-scale clinical trials of ABM for depression. Aim 1 is to conduct a randomized clinical trial among adults with elevated symptoms of depression and a negative attention bias that compares the efficacy of active ABM to cognitive control training and an assessment-only control condition that does not involve any ABM procedures. Aim 2 is to examine whether ABM alters negative attention bias and functional connectivity within frontal-parietal neural circuitry that support negative attention bias. Aim 3 is to identify mechanisms responsible for the putative efficacy of active ABM and cognitive control training. Study Impact: The current project proposes to target and reduce negative attention bias with a novel intervention grounded in basic psychopathology research. The investigators believe this experimental medicine approach will lead to the development of a highly specific and targeted intervention, using cutting-edge cognitive neuroscience to inform treatment development, and improve the quality of life of people whose psychopathology is maintained by negative attention bias.

ELIGIBILITY:
Inclusion Criteria:

* able and willing to provide informed consent;
* fluent in English;
* moderate or greater depression symptoms;
* attention bias for negative stimuli;
* stable psychiatric and neurological medication usage.

Exclusion Criteria:

* meets criteria for current substance use disorder (mild or greater severity), current or past psychotic disorder, bipolar disorder, or schizophrenia;
* has any medical or physical conditions that would preclude participation in an fMRI study (e.g., orthodontic braces);
* is currently receiving psychotherapy or electroconvulsive therapy (ECT);
* current opioid analgesics or systemic corticosteroid use for an acute medical condition or taken as needed;
* has had suicidal behaviors or significant suicidal ideation within the last six months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depression - Self Report (QIDS-SR) | Change in QIDS-SR from baseline to Week 4 to measure change in self-reported depression.
  16-item self-report measure of depression symptom severity

SECONDARY OUTCOMES:
Mood and Anxiety Symptoms Questionnaire-Short Form (MASQ-SF) | Change in MASQ-SF from baseline to Week 4 to measure change in self-reported depression.
  30-item self-report measure of negative affect symptoms
Hamilton Depression Rating Scale - 17 Item (HAMD-17) | Change in HAMD-17 from baseline to Week 4 to measure change in interviewer-rated depression.
  17-item clinician-administered measure of depression symptom severity

OTHER OUTCOMES:
Attention bias (eye tracking) | Change in attention bias from baseline to Week 4 to measure change in negative attention bias.
  Primary ABM treatment target
Resting State (fMRI) | Change in resting state fMRI from baseline to Week 4 to measure change connectivity in frontal-parietal brain circuitry.
  Resting state functional connectivity
Psychomotor vigilance test (PVT) | Change in PVT from baseline to Week 4 to measure change in sustained attention.
  Behavioral assessment of sustained attention

CONTACTS AND LOCATIONS:
Locations (1):
- Mood Disorders Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon study completion.

REFERENCES:
- [Result] Beevers CG, Clasen PC, Enock PM, Schnyer DM. Attention bias modification for major depressive disorder: Effects on attention bias, resting state connectivity, and symptom change. J Abnorm Psychol. 2015 Aug;124(3):463-75. doi: 10.1037/abn0000049. PMID 25894440
- [Derived] Beevers CG, Hsu KJ, Schnyer DM, Smits JAJ, Shumake J. Change in negative attention bias mediates the association between attention bias modification training and depression symptom improvement. J Consult Clin Psychol. 2021 Oct;89(10):816-829. doi: 10.1037/ccp0000683. PMID 34807657